CLINICAL TRIAL: NCT04085237
Title: The Benefit of Adding Ultrasound-guided ESP Block to PCA vs. PCA Alone for Postoperative Analgesia After Laparoscopic Nephrectomy Surgeries: a Pilot, Randomized Controlled Trial
Brief Title: ESP Block for Laparoscopic Nephrectomy Surgeries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was terminated because of poor recruitment rate.
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7119
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Kidney Cancer; Post-surgical Pain
MeSH Terms: conditions — Kidney Neoplasms; Pain, Postoperative | interventions — Ropivacaine; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research Pharmacy will provide randomization/allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided continuous ESP block with opioid PCA (Experimental): A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the T7/T8 spinous process. The patient's skin will be anesthetized with 2% lidocaine. A Contiplex Echo ultra 360 18G needle with 20G × 55 cm Contiplex Echo catheter will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of 0.375% ropivacaine with 5mcg/mL of epinephrine will be injected in 5-mL aliquots through the needle (maximum of 3mg/kg) followed by insertion of the echo catheter system under direct vision 2-3 cm beyond the needle tip.
  Interventions: Drug: Ropivacaine injection
- Ultrasound-guided sham block and catheter with opioid PCA (Sham Comparator): The exact same procedure as the experimental group will be followed, substituting saline for local anesthetic at the same amounts and rate. As with the ESP group, the patients will have PCA initiated postoperatively in the PACU at the same doses.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Ropivacaine injection — 30ml of 0.375% ropivacaine with 5mcg/ml of epinephrine will be injected into the fascial plane on the anterior spinae muscle.
  Other Names: Naropin
  Arms: Ultrasound-guided continuous ESP block with opioid PCA
Other: Sham — Saline will be used at the same amounts as the ropivacaine arm.
  Other Names: Placebo
  Arms: Ultrasound-guided sham block and catheter with opioid PCA

SUMMARY:
Nephrectomy (kidney removal) is one of the most common surgical procedures in urologic practice. Recent advances in laparoscopic (keyhole) procedures have resulted in a significant decrease in open nephrectomies. Most laparoscopic surgeries are performed through 3 to 4 small (1 to 1.5 cm) incisions; however, laparoscopic nephrectomies for cancer include one of the incisions being extended to 7 to 10 cm for kidney removal. Although pain after laparoscopic surgery is somewhat less than that after open surgery, it is still significant, and opioid consumption is similar. Opioids have been a mainstay for the treatment of post-operative pain, but they are associated with many adverse effects and a potential for long-term use. Thus, combining opioid analgesia with other forms of analgesia has the potential to reduce opioid use. Paravertebral nerve blocks, where local anesthetic is injected near the spinal nerves, have recently shown good pain control in patients undergoing thoracic and abdominal surgeries. However, this technique is technically challenging, time consuming, and has the risk of significant side effects. Fascial plane blocks are an alternative to paravertebral blocks. Fascial plane blocks, where local anesthetic is injected in areas further away from the spinal nerves, are easier to perform than paravertebral blocks, and have fewer associated risks. A recently described fascial plane block, the Erector Spinae Plane (ESP) block, has been shown to be effective in controlling pain in a variety of surgeries. However, currently, there is little information regarding its use in laparoscopic nephrectomy. We are proposing this pilot randomized control trial to look at the feasibility of completing a larger randomized control trial to evaluate ESP blockade in patients undergoing laparoscopic nephrectomy for cancer. We will also investigate total opioid consumption, and pain scores at rest and during movement.

DETAILED DESCRIPTION:
While post-operative pain seems to be slightly decreased compared to open nephrectomies, pain from laparoscopic nephrectomy is still significant and opioid consumption is similar.Adequate management of post-operative pain is imperative in early post-operative mobilization. ¬Although opioids have been a mainstay for the treatment of post-operative pain, other strategies should be considered as opioids are associated with adverse effects, the potential for long-term opioid use, and even death. There have been an increasing number of opioid related deaths with 2,066 apparent opioid-related deaths in Canada over the first half of 2018. With the need to address the worsening opioid crisis, it is essential that other non-opioid strategies are explored and considered. Multimodal anesthesia has been one effort to reduce opioid use post-operatively. Increasingly, the literature shows that peripheral nerve blocks reduce post-operative opioid consumption in a vast variety of surgeries.

Traditionally patients undergoing laparoscopic nephrectomy have opioid patient controlled analgesia pumps (PCAs) for post-operative pain control. PCA is widely recognized as an effective technique after laparoscopic nephrectomy to reduce pain scores. A meta-analysis of 49 articles showed PCA had better postoperative pain control than nurse administered analgesics over most time intervals with higher patient satisfaction. Complications of a PCA include respiratory depression, confusion or sedation, nausea, pruritus, ileus, and insufficient analgesia. Paravertebral blocks (PVB) have recently showed promise and increasing clinical uptake due to a growing use of ultrasound-guided regional anesthesia. They provide good pain control in patients undergoing thoracic and abdominal surgeries. In PVB, local anesthetic is injected near the thoracic spinal nerve at its exit from the intervertebral foramina, which results in unilateral somatic and sympathetic nerve blockade in multiple continuous thoracic dermatomes above and below the site of injection. However, this technique is technically challenging, time consuming, and carries a risk of pneumothorax. Fascial plane blocks are increasingly used as an alternative regional anesthetic strategy for abdominal surgery.

Recently ultrasound-guided Erector Spinae Plane (ESP) block was described in which local anesthetic is injected around the erector spinae muscle which tends to block the dorsal and ventral rami of the thoracic spinal nerves. There is growing evidence of its use in a wide range of surgeries. The appeal of the ESP block is in providing analgesia without the potential for needle pleura interaction and the consequent risk of pneumothorax. This interfascial block involves ultrasound guided injection of local anesthetics under the erector spinae muscle and superficial to transverse process of thoracic vertebrae at appropriate level. The ESP block targets the dorsal and ventral rami of the spinal nerves as they leave the intervertebral foramen. Cadaveric examination of ESP block showed extensive cranial-caudal spread of the block, approximately four dermatomes above and below the site of injection. The fact that the site of injection is distant from the spinal cord and pleura, increases the safety of the ESP block as compared to a paravertebral block. The transverse process is easily visualized on ultrasound and acts as a backstop for the needle, preventing excessively deep placement. Of importance, a catheter can also be placed easily during the ESP block allowing continuous infusion and prolonged analgesia. Given the importance of providing adequate analgesia in patients undergoing laparoscopic nephrectomy and the lack of consensus amongst surgeons and anesthesiologists for the optimal analgesic technique, we are proposing a pilot randomized controlled trial (RCT) to determine the feasibility of a larger RCT to compare continuous ESP blockade vs a Sham blockade. Both groups will receive opioid PCA and other multimodal analgesia combined with opioid PCA versus opioid PCA alone.

Literature review: We conducted a review via Pubmed looking at all studies associated with "erector spinae block". Of the studies found, 123 relevant studies were reviewed. The studies included 92 case reports and 4 randomized control trials, with the others being anatomical reviews, editorials, or small review articles. Of these, there were only 4 patients from 1 case series article where patients received ESP blocks for laparoscopic nephrectomies. None of these patients required post-operative opioids in addition to their ESP block infusions. We also reviewed clinicaltrials.gov for ongoing and proposed trials related to the ESP block. Currently, we identified 51 studies involving the ESP block. The vast majority of these revolved around thoracic and general surgery, including some randomized controlled trials. There was only 1 proposed trial studying the use of the ESP block with nephrectomies, but this one was evaluating surgeries

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring laparoscopic nephrectomy and partial nephrectomy for malignancy
* Patients of age 18 and over
* BMI < 40
* Patients who are expected to stay in-hospital overnight after surgery

Exclusion Criteria:

* Patient refusal
* Contraindications to paravertebral blocks: Infection at the site of needle insertion, empyema, allergy to local anesthetic drugs, and tumor occupying the thoracic paravertebral space, coagulopathy, bleeding disorder or therapeutic anticoagulation
* Known allergy to local anesthetics
* Inability to provide informed consent
* Inability to use a PCA due to languate or comprehension barriers
* BMI >= 40
* Any patient on opioids for greater than or equal to 3 months duration prior to surgery
* Patients with chronic pain syndromes
* Donor nephrectomies due to incision location
* Cystic kidney because of very large incisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Feasibility - Enrollment rate of greater than one patient per week with 100% in-hospital follow-up | One week
  Number of patients recruited per week

SECONDARY OUTCOMES:
Opioid Consumption | 48 hours
  Total long acting opioid consumption in hydromorphone equivalents
Pain scores at rest and movement | Day 1
  Pain scores will be recorded at intervals. The Numerical Rating Scale (NRS) is an 11-point scale where 0 is no pain and 10 is the worst pain imaginable.
Number of Adverse Events | Day 1-2
  Incidence of postoperative nausea-vomiting; respiratory depression; itching; local anesthetic toxicity; catheter leakage and catheter migration; infection at catheter site

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Lambe, MD, Principal Investigator — St. Joseph's Healthcare Hamilton and McMaster University; Peter Moisiuk, MD, Principal Investigator — St. Joseph's Healthcare Hamilton and McMaster University; Aaron Kugler, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Alper I, Yuksel E. Comparison of Acute and Chronic Pain after Open Nephrectomy versus Laparoscopic Nephrectomy: A Prospective Clinical Trial. Medicine (Baltimore). 2016 Apr;95(16):e3433. doi: 10.1097/MD.0000000000003433. PMID 27100439
- [Result] Shah A, Rowlands M, Krishnan N, Patel A, Ott-Young A. Thoracic Intercostal Nerve Blocks Reduce Opioid Consumption and Length of Stay in Patients Undergoing Implant-Based Breast Reconstruction. Plast Reconstr Surg. 2015 Nov;136(5):584e-591e. doi: 10.1097/PRS.0000000000001717. PMID 26505714
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016